CLINICAL TRIAL: NCT05622864
Title: Phase I Study on the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Single Dose Escalation of Nebulized Inhalation of HRS-9821 Suspension in Healthy Individuals and Multiple Doses in COPD Patients
Brief Title: Study on Single and Multiple Atomization Inhalation of HRS-9821 Suspension for Inhalation in Healthy Subjects and COPD Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRS-9821-I-101
Record Dates: First submitted 2022-11-14; First posted 2022-11-21 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental)
  Interventions: Drug: HRS-9821
- Part B (Experimental)
  Interventions: Drug: HRS-9821

INTERVENTIONS:
Drug: HRS-9821 — HRS-9821
  Arms: Part A
Drug: HRS-9821 — HRS-9821
  Arms: Part B

SUMMARY:
The increased safety and tolerance of single and multiple atomized inhalation of HRS-9821 suspension for inhalation doses in healthy subjects and COPD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an informed consent forms；
2. Healthy men aged 18-50 (both ends, subject to the signing of the informed consent form); COPD patients aged 40-75 (both ends, subject to the signing of the informed consent form);
3. Weight ≥45 kg，BMI 18-33 kg/m2 (include 33 kg/m2);
4. During the screening period, the vital signs of healthy subjects are normal:

   * Shrinkage 90-140 mmHg,
   * diastolic pressure 50-90 mmHg,
   * Heart rate 40-100 times/min;
5. During the screening period, the lung function of healthy subjects is normal, that is, the predicted value of FEV1≥80% and the predicted value of FEV1/FVC≥92%; After COPD patients inhale bronchodilators, he predicted value of FEV1≥40% and the predicted value of FEV1/FVC<0.7;
6. During screening, the 12-lead ECG is normal or abnormal but has no clinical significance.
7. Follow the contraceptive requirements within 14 weeks from the beginning of the consent to the last dose, and do not donate sperm during the consent period;
8. During the study, all research regulations and procedures can be followed, and the atomization devices used by the research institute can be used correctly;
9. Healthy subjects: non-smoking or quitting smoking ≥ 12 months, the previous smoking history < 5 packs of years; COPD patients: the previous smoking history ≥ 10 packs of years.

Exclusion Criteria:

1. Healthy subjects: in the past 12 weeks, antibiotics have been used for upper and lower respiratory tract infections, or have a history of respiratory infections within the past 4 weeks; COPD patients: in the past 4 weeks, antibiotics have been used for lower respiratory tract infections;
2. Healthy subjects: abnormal laboratory or physical examination results of clinical significance;
3. The average value of QTcF for 3 times at screening is ≥450ms;
4. In the past four weeks, there have been blood donations or large blood loss (more than 400 milliliters), or those who intentionally donate blood during the study;
5. Accept experimental drugs or use experimental medical devices within 1 months or less than 5 times the half-life of the drug, whichever is longer;
6. In the past, there were difficulties in collecting blood or could not withstand intravenous puncture, such as needle halo and blood halo
7. Any organ system has a history of malignant tumors;
8. Known to be allergic to any accessories in the research drug or formulation;
9. Previously known infection of human immunodeficiency virus (HIV), hepatitis B virus (HBV) liver or hepatitis C virus (HCV); or randomized pre-HIV (according to the test center SOP), treponema pallidum antibody (TPPA), HBV surface antigen or HCV antibody positive;
10. There is a history of smoking and alcoholism in the 3 months before screening: smoking (more than 5 cigarettes or equivalent tobacco per day); alcoholism (more than 14 units of alcohol per week: 1 unit = 360 mL of beer, or 25 mL of spirits with a concentration of 40% or more, or 1 glass of wine, 180mL);
11. In the past five years, there has been a history of drug abuse and drug dependence;
12. Before randomization, positive for alcohol or drug abuse or nicotine in urine;
13. During the study, there is a surgical plan or may interfere with the treatment plan carried out by the study;
14. Inability or unwillingness to fully comply with the research program;
15. Mentally or legally incapacitated;
16. The researchers believe that there are any other reasons why the subjects are unfit to participate in the study;
17. Prescription was used within 14 days before the first administration or within 48 hours before the first administration;
18. Drugs that have used strong/intermediate inhibitors or induce liver drug metabolic enzyme CYP3A4 14 days before the first administration or ingest grapefruit or related products within 7 days before the first administration;
19. During the study, it was expected to use drugs that had an effect on P-gp or breast cancer drug-resistant protein (BCRP).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Assess the incidence and severity of adverse events after single atomization inhalation of HRS-9821 in healthy subjects and multiple atomization inhalation of HRS-9821 in COPD patients. | About a month from the first medication to the evaluation.

SECONDARY OUTCOMES:
Evaluate the forced expiratory volume in one second (FEV1) after single atomization inhalation of HRS-9821 in healthy subjects and multiple atomization inhalation of HRS-9821 in COPD patients. | 2 hours after the first dose
Evaluate the forced expiratory volume in one second (FEV1) after single atomization inhalation of HRS-9821 in healthy subjects and multiple atomization inhalation of HRS-9821 in COPD patients. | 4 hours after the first dose
Evaluate the forced expiratory volume in one second (FEV1) after single atomization inhalation of HRS-9821 in healthy subjects and multiple atomization inhalation of HRS-9821 in COPD patients. | 6 hours after the first dose
Evaluate the forced expiratory volume in one second (FEV1) after single atomization inhalation of HRS-9821 in healthy subjects and multiple atomization inhalation of HRS-9821 in COPD patients. | 12 hours after the first dose
Evaluate the forced expiratory volume in one second (FEV1) after single atomization inhalation of HRS-9821 in healthy subjects and multiple atomization inhalation of HRS-9821 in COPD patients. | 24 hours after the first dose
Evaluate the average value of FEV1 compared with baseline changes after single atomization inhalation of HRS-9821 in healthy subjects and multiple atomization inhalation of HRS-9821 in COPD patients. | 2 hours after the first dose
Evaluate the average value of FEV1 compared with baseline changes after single atomization inhalation of HRS-9821 in healthy subjects and multiple atomization inhalation of HRS-9821 in COPD patients. | 3 hours after the first dose
Evaluate the average value of FEV1 compared with baseline changes after single atomization inhalation of HRS-9821 in healthy subjects and multiple atomization inhalation of HRS-9821 in COPD patients. | 4 hours after the first dose
Evaluate the average value of FEV1 compared with baseline changes after single atomization inhalation of HRS-9821 in healthy subjects and multiple atomization inhalation of HRS-9821 in COPD patients. | 12 hours after the first dose
Evaluate the average value of FEV1 compared with baseline changes after single atomization inhalation of HRS-9821 in healthy subjects and multiple atomization inhalation of HRS-9821 in COPD patients. | 24 hours after the first dose
Evaluate the change of FEV1 peak after single atomization inhalation of HRS-9821 in healthy subjects and multiple atomization inhalation of HRS-9821 in COPD patients. | About 24 hours after the first dose
Evaluate the force lung capacity (FVC) after single atomization inhalation of HRS-9821 in healthy subjects and multiple atomization inhalation of HRS-9821 in COPD patients. | 2 hours after the first dose
Evaluate pharmacokinetics concentration and pharmacokinetic parameters of after single atomization inhalation of HRS-9821 in healthy subjects and multiple atomization inhalation of HRS-9821 in COPD patients. | 2 weeks after the first dose

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital，Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided